CLINICAL TRIAL: NCT02134158
Title: Impact of Transcranial Direct Current Stimulation (tDCS) on Locomotion and Bipedal Equilibrium in Hemiplegic Patients: a Crossover Randomized Controlled Trial
Brief Title: Impact of tDCS on Locomotion and Equilibrium in Hemiplegic Patients
Acronym: HEMILOCOSTICOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P120135 / AOM12126; 2013-A00952-43 (Other: IDRCB)
Record Dates: First submitted 2013-12-18; First posted 2014-05-09 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Gait Disorders
Keywords: tDCS, gait disorders, equilibrium, hemiplegic, stroke
MeSH Terms: conditions — Mobility Limitation; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham and then anodal (Experimental): visit 2 sham stimulation (120 seconds) and visit 3 anodal stimulation (30 minutes)
  Interventions: Device: anodal tDCS and sham tDCS stimulations
- anodal and then sham (Experimental): visit 2 anodal stimulation (30 minutes) and visit 3 sham stimulation (120 seconds)
  Interventions: Device: anodal tDCS and sham tDCS stimulations

INTERVENTIONS:
Device: anodal tDCS and sham tDCS stimulations — Two conditions will be tested in randomized order: 2 arms in the first one anodal tDCS and then sham tDCS. In the other arm sham tDCS and then anodal tDCS.
  All the investigations will associate with clinical, functional and 3D motion analysis assessments.

SUMMARY:
The aim of this trial is to quantify the improvement of locomotion and equilibrium induced par tDCS in anode polarity position in post stroke hemiplegic patients.

DETAILED DESCRIPTION:
This is a pilot prospective randomised crossover double blind study. 40 patients will be enrolled in two sites, with 20 patients each site.

The duration of this study is planned to be 25 months: 24 months will be for enrollment and 1 month for the follow-up.

The follow-up of patient comprises 3 visits, will be extended to 28 days for each patient:

• V1: inclusion visit:

After obtained an informed consent signed, the following analysis will be realized: a clinical assessment, quantify analysis of walking using 3D motion analysis system, assessment of equilibrium using force plate and functional abilities.

The patient will record him-self clinical scales and will respond auto-evaluation questionnaires. A cerebral magnetic resonance imaging and a blood collection of 5 ml will also be realized.

• V2-V3 (Locomotion /equilibrium assessment visit):

V2 and V3 will begin with tDCS experimental visit (EV) or tDCS placebo visit (PV), the visit order for each patient will be defined by randomization result.

During the 2 visits, the tDCS will be placed on the scalp of the patient. The anode will be placed at the hot spot of the tibialis anterior motor cortex area on the damage hemisphere, and the cathode will be placed at the controlateral orbit. The intensity of stimulation will be 2 mA.

In tDCS experimental visit, the stimulation will last 30 minutes. In tDCS placebo visit, the duration of the stimulation will only be 120 seconds, with the identical other conditions.

Before the beginning of the stimulation, a clinical assessment, a functional gait related activities evaluation and a 3D gait motion analysis associated with an evaluation of the equilibrium will be performed.

During the stimulation period, the gait and the equilibrium assessments, using 3D motion analysis will be done.

After the stimulation, the evaluations such as clinical, functional and motion analysis will be realized again.

The tDCS experimental visit and the tDCS placebo visit will be spaced one week.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Unilateral stroke
* More than 6 months after stroke
* Ability to walk during 10 minutes without stopping
* Informed consent signed

Exclusion Criteria :

* Patient with pacemaker
* Claustrophobia (unable to perform a magnetic resonance imaging analysis)
* Patient with severe aphasia or severe cognitive disorder interfering the follow-up of the trial
* Neuro-orthopedic surgery history in the last 6 months on the studied paretic lower limb
* Epilepsy history in the last year
* Lack of medical insurance
* Adult patient under the care of a guardian
* Patient with progressive concomitant disease
* Patient with deep brain stimulation treatment (implantation of medical device)
* Patient with implantation of Intracranial metallic clip
* Patient with implantation of Intracranial stent
* Patient with implantation of ventriculoperitoneal derivation
* Patient with implantation of intracerebral or ocular prosthetic materials
* Patient with ferro-magnetic foreign object
* Patient with cochlear implant
* Patient with implantable cardioverter-defibrillator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Quantify of variability of the center-of-mass movement | 30 minutes
  Variability of the center-of-mass will be quantified during walking analysis and equilibrium assessment, for experimental and placebo visits (before, during and after stimulation) (V2 and V3) as well as in inclusion visit (V1).

SECONDARY OUTCOMES:
Symmetry index calculating | 30 Minutes
  Symmetry index of the spatio-temporal parameters of gait Calculating methods of the symmetry: using the robinson index
Continuous relative phase | 30 Minutes
  Assessment of the inter-segment coordination of the thigh-leg and leg-foot using the continuous relative phase.
Functional data | 30 minutes
  Time of climbing and descending 10 stairs of 11 cm Timed Up and Go test Box and Block Test

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD, PhD, Principal Investigator — Laboratory of Movement Analysis, Raymond Poincaré Hospital
Locations (1):
- Raymond Poincaré Hospital, Garches, Hauts-de-Seine, France

REFERENCES:
- [Derived] Geiger M, Supiot A, Zory R, Aegerter P, Pradon D, Roche N. The effect of transcranial direct current stimulation (tDCS) on locomotion and balance in patients with chronic stroke: study protocol for a randomised controlled trial. Trials. 2017 Oct 23;18(1):492. doi: 10.1186/s13063-017-2219-6. PMID 29061169